CLINICAL TRIAL: NCT05649111
Title: A Study of the Effect of Different Doses of Difluprednate Eye Drops on the Intraocular Pressure After Phacoemulsification
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Hashiem, Lecturer of ophthalmology ,ophthalmology consultant, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 50-11-16
Record Dates: First submitted 2022-11-25; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Uveitis, Anterior
MeSH Terms: conditions — Uveitis, Anterior

STUDY DESIGN:
Intervention Model Description: * Group A (FDA dose): will receive Difluprednate 4 times per day for 1 week, then twice per day for 1 week and then once per day for 5 days starting 24 hours after the operation
  * Group B will receive Difluprednate 3 times per day for 4 days, then twice per day for 4 days and then once per day for 4 days starting 4 hours after the operation
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): will receive Difluprednate 4 times per day for 1 week, then twice per day for 1 week and then once per day for 5 days starting 24 hours after the operation
  Interventions: Drug: Difluprednate Eye Drops
- Group B (Active Comparator): will receive Difluprednate 3 times per day for 4 days, then twice per day for 4 days and then once per day for 4 days starting 4 hours after the operation
  Interventions: Drug: Difluprednate Eye Drops

INTERVENTIONS:
Drug: Difluprednate Eye Drops — post-operative cataract surgery medication regimen. but different dosages between the 2 groups.

SUMMARY:
The study aims at detecting the minimum effective daily dose and duration of difluprednate that can be used to treat postoperative inflammation after phacoemulsification without increasing the intraocular pressure, and whether it can be safely given within the first 24 hours after the operation.

DETAILED DESCRIPTION:
Conventional phacoemulsification will be performed by the same surgeon for all the cases using the stop and chop technique. Anterior chamber examination for flare and cells using slit-lamp biomicroscopy according to the SUN recommendations and intraocular pressure measurement using Goldmann applanation tonometer will be done for all the cases before surgery and on the 1st, 3rd, 7th, 14th days as well as one month after the procedure.

All cases will receive Nepafenac 0.1% ( Nevanac 0.1%) 3 times per day on the last preoperative day, one tablet of Acetazolamide 250 mg (Cidamex 250mg) within the first 3 hours after the procedure and Moxifloxacin (Vigamox 0.5%) 0.1 ml intracameral and post-operative drops 3 times per day for 10 days and will be divided into:

In this pilot study:

* Group A : will receive Difluprednate 4 times per day for 1 week, then twice per day for 1 week and then once per day for 5 days starting 24 hours after the operation
* Group B : will receive Difluprednate 3 times per day for 4 days, then twice per day for 4 days and then once per day for 4 days starting 4 hours after the operation

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80
* Grade 1 to 4 nuclear cataract LOCS II
* Cumulative dissipated energy CDE 1 to 10
* Done by a single surgeon using the chopping technique

Exclusion Criteria:

* History of uveitis
* the use of topical or systemic steroids on the last post-operative day
* Intraoperative or postoperative complications
* Intraoperative iris manipulations or phaco traume

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Anterior chamber examination for flare and cell | 3 months
  using SUN classification

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hashem, PhD, Principal Investigator — Kafrelsheikh university faculty of medicin
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No